CLINICAL TRIAL: NCT05371691
Title: A Comparison of the Effectiveness of Two Types of Myofunctional Appliances: A Randomized Clinical Trial
Brief Title: A Comparison of the Effectiveness of Two Types of Myofunctional Appliances
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Mushriq F. Abid, Professor, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 387421
Record Dates: First submitted 2022-04-26; First posted 2022-05-12 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Tooth Position Anomalies
Keywords: Myofunctional appliance; Myobrace.; Twin-block; Cl II div I malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding to treatment allocation is possible only for the outcomes assessor because the clinicians could know the intervention. All the trial documents will be labeled with the study ID number, which be used for participant identification and data collection without unmasking the allocation group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myobrace group (Experimental): Myobrace appliance will be used for children who have Cl.II div.a malocclusion
  Interventions: Device: Myofunctional appliance
- Twin-block group (Experimental): Twin-block appliance will be used for children who have Cl.II div.a malocclusion
  Interventions: Device: Myofunctional appliance

INTERVENTIONS:
Device: Myofunctional appliance — Myifunctional appliance will be used for growing patients who have Cl.II div.1 malocclusion, two types of appliances are involved myobrace and twin=block appliance

SUMMARY:
A randomized clinical trial is set out to compare the effectiveness of two types of functional appliances in the correction of a Class II malocclusion. (Class II malocclusions are where upper front teeth bite significantly further forward in relation to lower front teeth).

DETAILED DESCRIPTION:
It is a multicenter randomized clinical trial with two arms parallel group. The patients will be randomly divided into two groups, group one: Myobrace appliance will be used while, and group two Twin-block appliances will be used. Cephalometric x-ray will be taken before starting the treatment (T1) and at the end of treatment (T2) at 9 months. The effectiveness of the two appliances will be assessed and measured comparing the difference in the cephalometric X-ray before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Growing children who need myofunctional appliance.
2. Cl II div. 1 malocclusion.
3. No previous orthodontic or orthopaedic treatments.

Exclusion Criteria:

1. Patients with systemic involvement.
2. Congenital malformations such as cleft lip and palate.
3. Facial deformities.
4. Finger sucking habit will be excluded

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
Dentoskeletal changes | T1 at the start of treatment and T2 at the end of treatment around 9 months
  Evaluation of dentoskeletal and soft tissue changes following the treatment of growing children with myobrace and twin block appliances. Using cephalometric analysis to measure the angles including dental angles such as inter-incisal angle, in addition to skeletal angles such as SNA,SNB and ANB angles.

SECONDARY OUTCOMES:
Soft tissue changes | T1 at the start of treatment and T2 at the end of treatment around 9 months
  2. Soft tissue changes using cephalometric radiographs including different angular measurement such as E-line and nasolabial angle (comparing the changes in the photographs at the beginning of the treatment and at the end of the treatment.
Patient satisfaction | At the end of treatment (around 9 months)
  3.Patient satisfaction with both appliances will be investigated using a questionnaire at the end of the study (around 9 months)

CONTACTS AND LOCATIONS:
Locations (2):
- Iraq (2):
  - College of Dentistry-University of Baghdad, Baghdad, Al-Rusafa
  - College of Dentisry-University of Baghdad, Baghdad